CLINICAL TRIAL: NCT02838368
Title: Investigating Pompe Prevalence in Neuromuscular Medicine Academic Practices
Acronym: IPANEMA
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Tahseen Mozaffar, Professor, University of California, Irvine
Other Study IDs: UCI-Ipanema
Record Dates: First submitted 2016-05-12; First posted 2016-07-20 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2018-08

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The incidence of type II glycogen-storage disease (Pompe disease) varies depending on ethnicity and geographic region. As of 2010, nine studies have been published documenting the incidence of Pompe disease. It is most common within the African American population, with an incidence of 1 in 14,000. In the U.S. more broadly speaking, the combined incidence of all three variants of the disease is 1 in 40,000. These estimates relied on the frequencies of three mutations in the gene acid alpha-glucosidase (GAA), leading to variants of the disease. Criteria for inclusion in the studies were often non-selective; in many cases, molecular genetic screening was done at birth. With such a high prevalence of Pompe disease reported, it is expected that large university medical centers specializing in neuromuscular diseases would see a higher incidence of Pompe disease among their patients. From a comparable Italian multicenter study, it appears that Pompe disease accounts for 3% of all patients presenting with proximal weakness with or without CK elevation.

This study will measure the incidence of Pompe disease based on manifest laboratory abnormality, namely low GAA enzyme activity. Analysis of GAA enzyme activity will be determined through a blood sample of 4 mL. The study seeks to measure the epidemiology of Pompe disease by symptomatically screening all patients who present with symptoms of hitherto undiagnosed proximal weakness with or without elevation of the muscle enzyme, creatinine kinase (CK), or elevation of CK alone, at thirteen academic tertiary neuromuscular practices throughout the United States and Canada. Total recruitment is expected to be ~1,500 participants. It is anticipated that the number of incident Pompe cases in this cohort would be between 3-5%, i.e. 45-75 newly diagnosed cases of Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 years or older.
* Geographically accessible to one of the sites.
* One of these following three clinical situations: Complaint of proximal muscle weakness with or without elevation in creatinine kinase (CK); neck muscle weakness (either flexor or extensor) with or without elevation in CK; or elevation of CK in isolation.
* Capable and willing to provide informed consent or assent and follow study procedures.

Exclusion Criteria:

* Less than 8 years of age.
* Subjects with an alternative neuromuscular diagnosis that is responsible for subject's symptoms
* Incapable or unwilling to provide informed consent and to follow research procedures.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients age of 8 years and older suspected of late-onset Pompe disease.
Sampling Method: Probability Sample
Enrollment: 921 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The true incidence of Pompe disease among patients seen at neuromuscular clinics. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Tahseen Mozaffar, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

REFERENCES:
- [Background] Cupler EJ, Berger KI, Leshner RT, Wolfe GI, Han JJ, Barohn RJ, Kissel JT; AANEM Consensus Committee on Late-onset Pompe Disease. Consensus treatment recommendations for late-onset Pompe disease. Muscle Nerve. 2012 Mar;45(3):319-33. doi: 10.1002/mus.22329. Epub 2011 Dec 15. PMID 22173792
- [Background] Sperry E, Leslie N, Berry L, Pena L. Pompe Disease. 2007 Aug 31 [updated 2025 Aug 21]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1261/ PMID 20301438
- [Background] Hirschhorn R, Reuser AJ. Glycogen storage disease type II: acid alpha-glucosidase (acid maltase) deficiency. In: Scriver CR, Beaudet A, Sly WS, Valle D, eds. The Metabolic and Molecular Bases of Inherited Disease. New York, NY: McGraw-Hill; 2001:3389-420.
- [Background] Martiniuk F, Chen A, Mack A, Arvanitopoulos E, Chen Y, Rom WN, Codd WJ, Hanna B, Alcabes P, Raben N, Plotz P. Carrier frequency for glycogen storage disease type II in New York and estimates of affected individuals born with the disease. Am J Med Genet. 1998 Aug 27;79(1):69-72. doi: 10.1002/(sici)1096-8628(19980827)79:13.0.co;2-k. No abstract available. PMID 9738873
- [Background] Musumeci O, la Marca G, Spada M, Mondello S, Danesino C, Comi GP, Pegoraro E, Antonini G, Marrosu G, Liguori R, Morandi L, Moggio M, Massa R, Ravaglia S, Di Muzio A, Filosto M, Tonin P, Di Iorio G, Servidei S, Siciliano G, Angelini C, Mongini T, Toscano A; Italian GSD II group. LOPED study: looking for an early diagnosis in a late-onset Pompe disease high-risk population. J Neurol Neurosurg Psychiatry. 2016 Jan;87(1):5-11. doi: 10.1136/jnnp-2014-310164. Epub 2015 Mar 17. PMID 25783438
- [Derived] Wencel M, Shaibani A, Goyal NA, Dimachkie MM, Trivedi J, Johnson NE, Gutmann L, Wicklund MP, Bandyopadhay S, Genge AL, Freimer ML, Goyal N, Pestronk A, Florence J, Karam C, Ralph JW, Rasheed Z, Hays M, Hopkins S, Mozaffar T. Investigating Late-Onset Pompe Prevalence in Neuromuscular Medicine Academic Practices: The IPaNeMA Study. Neurol Genet. 2021 Oct 18;7(6):e623. doi: 10.1212/NXG.0000000000000623. eCollection 2021 Dec. PMID 36299500